CLINICAL TRIAL: NCT02515487
Title: An Investigation of Chemotherapy Induced Cognitive Impairments in Breast Cancer
Brief Title: An Investigation of Chemotherapy Induced Cognitive Impairments in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-00146
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Post-chemotherapy; cognitive impairment
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients receiving chemotherapy treatment (Experimental)
  Interventions: Other: Brain Fitness Program (BFP)

INTERVENTIONS:
Other: Brain Fitness Program (BFP) — The program is designed to improve processing speed of auditory information and attention. The BFP is comprised of six computerized subtests that continuously adjust in the level of difficulty to maintain an 85% correct response rate. The subtest exercises include discrimination of confusable syllables, recognition of sequences of syllables, matching pairs of confusable syllables, reconstruction of sequences of verbal instructions and identification of details in a verbally presented story. Participants will participate in 40 one-hour training sessions over a 12 week period to complete all cognitive remediation training sessions. Since this intervention is presented both visually and verbally, noise cancelling headphones will be provided to the participants.

SUMMARY:
The main goal of this project is to identify and remediate the cognitive difficulties, including processing speed and attention deficits in individuals who have undergone chemotherapy treatment. Recent research has demonstrated objective cognitive deficits following chemotherapy and that it is not an emotional reaction to the cancer diagnosis as it was once considered. There are a large number of woman diagnosed and treated for breast cancer that experience chemotherapy induced cognitive deficits.

Subjects who participate in the study will be evaluated for cognitive abilities prior to chemotherapy treatment and after completion of chemotherapy. Participants will then have the option to participate in the second phase of the study, which involves the use of a computer-based Brain Fitness Program for 12 weeks. This is followed by another cognitive evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast cancer with adjuvant chemotherapy treatment
2. all subjects will be between the ages of 18 and 70 years old
3. free from significant psychiatric history
4. free of current alcohol or drug abuse.
5. All participants need to understand and read English and have the capacity to consent.

Exclusion Criteria:

1. Individuals with pre-exiting neurological disorder (i.e. brain tumors, dementia, Parkinson's disease, multiple sclerosis, seizure disorder) or diagnosed with metastasis cancer.
2. Individuals younger than 18 years old and older than 70 years old will also be excluded due to developmental changes that occur in those years.
3. Individuals with a current substance use disorder will also be excluded.
4. Individuals who lack the capacity to consent will be excluded from this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Wechsler Test of Adult Reading (WTAR) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  The WTAR is a measure that reliably estimates levels of intelligence by asking the subject to read aloud the words on an established reading list.
Change in Processing Speed (PS) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  1) The Paced Auditory Serial Addition Test (PASAT), which assesses complex mental manipulation of verbally presented single digit numbers. The task requires the participant to mentally add and verbally express the last two numbers presented. There are 60 trials in each of the two sets of numbers that are presented at two different speeds; 2) Symbol-Digit Modality Test requires that the subject copies numbers that are paired with symbols within a specified time limit. The coding subtest involves processing speed, short term visual memory, psychomotor speed, visual perception and visual scanning ability. 3) The Stroop Test has three parts to it: the first task requires the participant to respond to every word as quickly as possible that is presented on the computer screen. The second task requires a response when the color word matches the meaning of the word. The third task requires a response when the color of the word does not match the meaning of the word.
Change in Executive Functions | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  The Trail Making Test, Part A & B: are measures of visual search efficiency and set shifting while alternating between letters and numbers. Additionally, the Verbal Fluency subtest of the Delis-Kaplan Executive Functioning Scale (D-KEFS) will be used to measure semantic and phonemic fluency through a task of word naming, where subjects are asked to list as many words as they can within 60-second time limit that begin with a specific letter (i.e., F, A, and S), and a task of category naming, where subjects are asked to list as many words as they can within 60-second time limit that fall within a specified category (i.e., animals and boy's names), respectfully. This subtest also measures category switching ability via a task where subjects are asked to list as many words as they can within 60-second time that fall within two alternating categories (i.e., fruits/furniture).
Change in Working Memory and Attention | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  1) Digit-Span Task, this is a standardized measure of verbal working memory in which participants recall a string of numbers that are verbally presented. 2) The Continuous Performance subtest of the CNS Vital Signs neurocognitive battery. The Continuous Performance test assesses sustained attention and reaction time to targets presented on the computer by requiring the participant to respond only when a specific designated letter is presented during a 5 minute trial. 3) The Shifting Attention subtest of the CNS- Vital Signs neurocognitive battery will be administered to assess the participant's ability to maintain attention while switching between sets of target. 4) Four-Parts Continuous performance subtest of the CNS Vital Signs neurocognitive battery, which is a measure of working memory and sustained attention.
Change in Visual and Verbal Memory | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  Verbal memory will be assessed with the California Verbal Learning Test (CVLT-II) which assesses learning and rote memory of verbal material. Subjects are verbally presented with a list of words that are assessed immediately and after a 20-minute delay with and without cues. The short form version of this test will be used. The Visual Memory subtest of the CNS- Vital Signs neurocognitive battery will be administered to assess non-verbal memory of immediate and delayed recall.
Change in Depression | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  Beck Depression Inventory -II: This is a standardized instrument for the assessment of depression with a self-report questionnaire. Participants will endorse the level of disturbance which best describe their mood over 21 items that are characteristic of depression.
Change in Anxiety | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  Beck Anxiety Inventory (BAI): The BAI is a self-report instrument for the assessment of anxiety. The BAI consists of 21 items, each describing a common symptom of anxiety on which the respondent rates how much they have been bothered by the symptoms over the last week.
Change in Frontal Systems Behavior Scale (FRSBE) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  A validated self-report of three frontal systems behavioral syndromes: apathy, disinhibition, and executive dysfunction.
Change in Cognitive Self-Report Questionnaire (CSRQ) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  A validated self-report questionnaire that assesses perceptions of cognition and mood related to everyday experiences for the past two weeks
Change in Functional Assessment of Cancer Therapy-Cognitive Scale (FACT-Cog) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  Measures patient's perceived cognitive functioning as a result of their diagnosis and cancer therapy.
Change in Functional Assessment of Cancer Therapy - Fatigue scale (FACIT-F) | Difference from baseline to end of chemotherapy (approximately 4 months, depending on individual treatment); difference from end of chemotherapy to 12 weeks post-chemotherapy
  A measure of one's perception of their level of Fatigue as a result to cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Voelbel, PhD, Principal Investigator — New York University
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States